CLINICAL TRIAL: NCT02371018
Title: Acute Effects of Nutrition Supplementation on Treatment Efficiency and Hemodynamics During Dialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 14385
Record Dates: First submitted 2015-02-05; First posted 2015-02-25 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2017-09

CONDITIONS: Blood Pressure; Kidney Failure, Chronic; Dietary Modification
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard Hemodialysis (No Intervention): Participants will be monitored during their normal hemodialysis treatment with no intervention administered
- Hemodialysis with Nutrition Supplement (Experimental): Participants will be monitored during a normal hemodialysis treatment in which they consume 1-8oz can of Nepro.
  Interventions: Dietary Supplement: Nepro
- Nutrition Supplement (Experimental): Participants will be monitored while drinking 1-8oz can of Nepro with no hemodialysis treatment.
  Interventions: Dietary Supplement: Nepro

INTERVENTIONS:
Dietary Supplement: Nepro — Patients will be asked to consume a single 8 oz can of Nepro
  Arms: Hemodialysis with Nutrition Supplement; Nutrition Supplement

SUMMARY:
The purpose of this study is to examine the effect of nutritional supplementation during hemodialysis treatment on beat-to-beat hemodynamics and treatment efficiency in a crossover design.

DETAILED DESCRIPTION:
The consumption of food or nutritional supplements during hemodialysis treatment has been shown to improve nutritional status, improve quality of life, and reduce mortality.

Despite these observations, allowing patients to eat food during hemodialysis treatment is sometimes restricted in the United States. The reasons for this restrictive policy are multi-factorial, but include concerns related to drops in blood pressure BP or a reduced efficiency of solute removal following eating during HD treatment. An alternative to eating solid food is to provide patients with liquid nutritional supplements. Clinics in the US are more likely to allow the consumption of liquid nutritional supplements, however, little is known about the effect that liquid supplements have on blood pressure or treatment efficiency. Therefore, the investigators plan to examine the effect of nutritional supplementation during hemodialysis treatment on hemodynamics and treatment efficiency in a crossover design.

ELIGIBILITY:
Inclusion Criteria:

* Receiving hemodialysis treatment three times per week, on hemodialysis for greater than three months, receive medical clearance from a Nephrologists

Exclusion Criteria:

* Milk or soy allergy, more than 4 hypotensive events requiring intervention in the last two weeks, hospitalized due to hypotension in the previous week

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-02 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Changes in beat-to-beat systolic blood pressure | Duration of each treatment (approximately four hours), treatments will be one week apart for a total of three weeks
  Beat-to-beat blood pressure will be monitored throughout the treatment by finger plethysmography

SECONDARY OUTCOMES:
Gastrointestinal symptoms during treatment by a rating scale | Duration of each treatment (approximately four hours), treatments will be one week apart for a total of three weeks
  A validated version of the Gastrointestinal Symptom Rating Scale will be administered
Treatment efficiency measured by urea removal | Duration of each treatment (approximately four hours), treatments will be one week apart for a total of three weeks
  Kt/V as determined from blood urea pre- and post-hemodialysis

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth R Wilund, PhD, Principal Investigator — University of Illinois at Urbana-Champaign
Locations (1):
- University of Illinois, Urbana, Illinois, United States

REFERENCES:
- [Derived] Mah JY, Choy SW, Roberts MA, Desai AM, Corken M, Gwini SM, McMahon LP. Oral protein-based supplements versus placebo or no treatment for people with chronic kidney disease requiring dialysis. Cochrane Database Syst Rev. 2020 May 11;5(5):CD012616. doi: 10.1002/14651858.CD012616.pub2. PMID 32390133